CLINICAL TRIAL: NCT00575809
Title: Incidence and Factors Associated With the Development and Severity of Oral Mucositis in Patients Undergoing High-Dose Chemotherapy and Peripheral Blood Stem Cell Transplantation
Brief Title: Incidence and Factors Associated With the Development and Severity of Oral Mucositis
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: South Texas Veterans Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: HSC20050218H
Record Dates: First submitted 2007-12-15; First posted 2007-12-18 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Peripheral Blood Stem Cell Transplantation
Keywords: Mucositis, hematopoietic stem cell transplantation, chemotherapy
MeSH Terms: conditions — Mucositis | interventions — Nutrition Assessment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obsevational
  Interventions: Other: Mucositis and nutritional assessments

INTERVENTIONS:
Other: Mucositis and nutritional assessments — Mucositis and nutritional assessments before and during the hematopoietic stem cell transplantation

SUMMARY:
Our study intends to evaluate prospectively the incidence and severity of oral mucositis in patients undergoing high-dose chemotherapy and hematopoietic stem cell transplantation, as well as to evaluate the potential influence of nutritional-, physical-, and transplant-related factors associated with the development of this complication and its grade of involvement.

DETAILED DESCRIPTION:
Objective: Our study intends to evaluate prospectively the incidence and severity of oral mucositis in patients undergoing high-dose chemotherapy and hematopoietic stem cell transplantation, as well as to evaluate the potential influence of nutritional-, physical-, and transplant-related factors associated with the development of this complication and its grade of involvement.

Research plan: This is a prospective cohort study with an observational basis that involves all of the patients undergoing high-dose chemotherapy and peripheral blood stem cell transplantation at the Audie L. Murphy VA Hospital Bone Marrow Transplant Unit and at the University Hospital Bone Marrow Transplant Unit. We expect to enroll 400 patients during a 5-year period.

Methods: In order to answer the study questions, subjects will be assessed several times during the study period. The study involves a multidisciplinary group that will be evaluating and following the subjects. A baseline will be established by a physician and a nutritionist before the subjects start the high-dose chemotherapy regimen. The subjects will be followed with oral evaluations 3 times per week, beginning on the day of the transplant and ending when mucositis resolves, or the patient is discharged home, or 30 days post-transplant, whichever occurs first. At day 15 post-transplant, patients will be evaluated for the second time by the nutritionist. Further information such as blood values, use of medications and treatment complications, will be obtained by daily chart review.

Clinical relevance: Mucositis is, without a doubt, one of the most common and debilitating complications resulting from the intense cytotoxic therapies preceding hematopoietic stem cell transplantation. Mucositis is not only a problem for the patient who needs to deal with the pain and the rapidly decreasing quality of life, but it is also a problem for the health system. Mucositis frequently results in increased hospital length of stay, resulting in a significant increase in the cost of medical care. Multiple prophylactic and therapeutic attempts have been made in order to control the symptoms and the severity of mucositis. No prevention or cure is available for the disease. Despite the renewed interest in this complication, important gaps in knowledge remain in this area of the supportive care of cancer patients. These gaps in knowledge are wider in the area of mucositis in patients who undergo hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hematopoietic stem cell transplantation
* Age 18 years and older
* Patients must understand and sign the study informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing hematopoietic stem cell transplantation
Sampling Method: Non-Probability Sample
Enrollment: 633 (Actual)
Dates: Start 2005-05; Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
To evaluate the incidence and severity of oral mucositis in patients undergoing high-dose chemotherapy and hematopoietic stem cell transplantation | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Cesar O Freytes, MD, Principal Investigator — South Texas Veterans Health Care System
Locations (2):
- United States (2):
  - Department of Veterans Affairs, South Texas Veterans Health Care System, Audie L. Murphy Memorial Veterans Hospital Division, San Antonio, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas